CLINICAL TRIAL: NCT01944670
Title: Multi-Center Trial to Evaluate an Internal Joint Stabilizer - Elbow ("IJS-E")
Brief Title: Multi-Center Trial to Evaluate an Internal Joint Stabilizer - Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skeletal Dynamics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLP-00015-00RAA
Record Dates: First submitted 2013-09-10; First posted 2013-09-18 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Trauma; Chronic Elbow Dislocation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Internal Joint Stabilizer Group (Experimental): Patients implanted with the Internal Joint Stabilizer - Elbow (IJS-E)
  Interventions: Device: Internal Joint Stabilizer - Elbow (IJS-E)

INTERVENTIONS:
Device: Internal Joint Stabilizer - Elbow (IJS-E) — Device designed for internal stabilization of the elbow

SUMMARY:
The purpose of this study is to confirm the safety and effectiveness of the Internal Joint Stabilizer - Elbow.

ELIGIBILITY:
Inclusion Criteria:

* The subject is >21 years of age.
* The subject is considered a candidate for the Internal Joint Stabilizer -Elbow (IJS-E) under one of the following indications:

  * Subjects where either the elbow sublocates or dislocates after repairing the injured ligaments and/or bones
  * The elbow has been subluxated or dislocated for more than 10 days prior to surgery
  * The elbow subluxes or dislocates after surgical repair/reconstruction
* The subject has sufficient quantity or quality of bone. Specifically there is sufficient trochlea of the distal humerus and of sufficient quality that the axis pin of the IJS-E has a secure hold as judged by the surgeon intra-operatively. Also, the screws placed in the ulna must be judged by the surgeon to have sufficient hold.
* The subject or legal guardian has been informed of the nature of the study, agrees to its provisions, and has provided informed written consent.
* The subject is willing to be available for the appropriate follow-up for the duration of the study.

Exclusion Criteria:

* The subject has one of the following conditions:

  * Presents with limited elbow motion as opposed to instability (subjects where instability is created through surgical release for chronic limitation of movement, soft tissue release, removal of adhesions and heterotopic ossification and/or fascial interposition will be excluded).
  * Active infection, suspicion of colonization or quiescent infection
  * Bacteremia
  * Bone loss greater than 30% of the total articulation or involving an entire column of the distal humerus
  * The subject has less than 50% of the height of the coronoid remaining, based on lateral x-ray view
  * Osteoporosis to the degree that the screws that insert into the ulna loosen during implantation
  * Material sensitivity to titanium or cobalt chrome
* The subject has imminent, known issues related to life expectancy.
* The subject is unable and/or unwilling to cooperate with study procedures, a rehabilitative program, or required follow-up visits.
* The subject has a condition that may interfere with the outcome or impede healing.
* The subject, in the opinion of the Clinical Investigator, has an existing condition that indicates he/she is not a good candidate for the study.
* The subject is unable or unwilling to give informed consent and/or who has no responsible family member willing to give consent.
* The subject is transient and has no fixed address.
* The subject is a prisoner.
* The subject is <21 years of age, or >21 years of age but skeletally immature.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Internal Joint Stabilizer Group
Started | 26
Completed | 24
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Patients implanted with the Internal Joint Stabilizer - Elbow (IJS-E)
Arm/Group | Internal Joint Stabilizer Group
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height (in) [Mean (Standard Deviation); unit: inches] | 65.8 (4.0)
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 188.0 (41.2)
Side Dominance [Count of Participants; unit: Participants]
  Right Handed | 24
  Left Handed | 1
  Ambidextrous | 1
Operative Side [Count of Participants; unit: Participants]
  Dominant Hand (including ambidextrous patients) | 9
  Non-dominant Hand | 17
Subluxed or Dislocated [Count of Participants; unit: Participants]
  Subluxed | 7
  Dislocated | 19

OUTCOME MEASURES:

1. Primary Outcome: Broberg Morrey Functional Rating
Description: To confirm that the Internal Joint Stabilizer - Elbow (IJS-E) provides temporary stabilization of the elbow joint and allows functional recovery after trauma or chronic dislocation.
  The study is deemed a success if the at least 75% of patients receive a Broberg Morrey Functinoal Rating of Fair or better.
Time Frame: Eight months (6 months post-explant)
Population: Patients implanted with the Internal Joint Stabilizer - Elbow (IJS-E) who completed the study (have final follow-up data). Excludes patients who were lost to follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Completed the Study: Patients implanted with the Internal Joint Stabilizer - Elbow (IJS-E) who completed the study (have final follow-up data)
  Internal Joint Stabilizer - Elbow (IJS-E): Device designed for internal stabilization of the elbow
Arm/Group | Participants Who Completed the Study
Number analyzed (Participants) | 24
Participants
  Broberg Morrey Score of Excellent | 14
  Broberg Morrey Score of Good | 8
  Broberg Morrey Score of Fair | 1
  Broberg Morrey Score of Poor | 1

2. Primary Outcome: Recurrent Dislocations
Description: To confirm that the Internal Joint Stabilizer - Elbow (IJS-E) provides temporary stabilization of the elbow joint and allows functional recovery after trauma or chronic dislocation.
  The study is deemed a success if the at least 75% of patients do not have a recurrent dislocation while using the IJS-E or after removal of the IJS-E.
Time Frame: 8 months (6 month post-explant)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Completed the Study
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Arm/Group | Participants Who Completed the Study
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Who Completed the Study (N=24)
Inflammation (Infections and infestations) | 1 — Inflammation was observed at the explant site 10 days after the implantation in one patient. The surrounding tissue was cultured negative for infection, but the subject was treated with antibiotics as a precaution.

LIMITATIONS AND CAVEATS:
Two patients were lost to follow-up prior to IJS-E implant removal (explant).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No